CLINICAL TRIAL: NCT03378570
Title: The Effects of Repetitive Transcranial Magnetic Stimulation Prefrontal Target Location on Outcomes for Major Depressive Disorder
Brief Title: rTMS for MDD: 5.5cm Rule vs. F3 Targeting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nicholas Trapp (Other)
Responsible Party: Sponsor-Investigator, Nicholas Trapp, Physician-Associate and Neuromodulation Fellow, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201709834
Record Dates: First submitted 2017-12-14; First posted 2017-12-20 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Major Depressive Disorder; Depression
Keywords: Transcranial Magnetic Stimulation; rTMS; F3; 5.5cm rule; Targeting; TMS
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- 5.5cm Rule Group (Active Comparator): rTMS will be targeted at a left prefrontal target 5.5cm anterior to the primary motor strip identified on the scalp during motor threshold testing.
  Interventions: Device: Repetitive transcranial magnetic stimulation
- F3 Group (Active Comparator): rTMS will be targeted at the left prefrontal scalp target identified as F3 according to the 10-20 EEG system.
  Interventions: Device: Repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation — Repetitive transcranial magnetic stimulation will be targeted to a location in the left prefrontal cortex and delivered according to FDA-approved parameters for the treatment of major depressive disorder, specifically high-frequency 10 Hz rTMS for 3000 pulses, 5 days per week for a total number of sessions as deemed clinically appropriate by the patient's clinical TMS treatment team but usually on the order of 20-30 treatments.

SUMMARY:
The purpose of this study is to examine the effects of different treatment locations using repetitive transcranial magnetic stimulation (rTMS) to treat major depressive disorder.

DETAILED DESCRIPTION:
Currently there is little standardization between rTMS treatment programs as to what is the best way to localize the left dorsolateral prefrontal cortex, which is the FDA-approved treatment location for clinical rTMS for major depressive disorder (MDD). Different targeting methods yield locations that can vary by up to a few centimeters. By comparing different treatment locations and obtaining neurobehavioral, neuroimaging, cognitive, and neuropsychological measures, this study would provide the opportunity to identify the optimal treatment targeting method when using rTMS for major depressive disorder in a clinical setting. This study will specifically be focusing on comparing the two most common targeting methods: a target 5.5cm anterior to the motor strip on the left prefrontal scalp and the F3 target location on the left prefrontal scalp as identified using the 10-20 EEG system nomenclature.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of major depressive disorder
* Age between 18 and 90 years
* rTMS is clinically indicated as determined by clinical rTMS physician team at University of Iowa

Exclusion Criteria:

* rTMS contraindication such as implanted ferromagnetic material in the head or history of epilepsy with poorly controlled seizures
* MRI exclusion criteria (if participating in MRI portion of study) including implanted device such as:
* Pacemaker
* Coronary Stent
* Defibrillator
* Neurostimulation
* Or any of the following conditions:
* Claustrophobia
* Uncontrolled high blood pressure
* Poorly controlled atrial fibrillation
* Significant heart disease
* Hemodynamic instability
* Severe kidney disease
* Pregnant, trying to become pregnant, or breast feeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-09-13 (Actual); Study Completion 2022-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas T Trapp, M.D., Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals & Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Trapp NT, Pace BD, Neisewander B, Ten Eyck P, Boes AD. A randomized trial comparing beam F3 and 5.5 cm targeting in rTMS treatment of depression demonstrates similar effectiveness. Brain Stimul. 2023 Sep-Oct;16(5):1392-1400. doi: 10.1016/j.brs.2023.09.006. Epub 2023 Sep 14. PMID 37714408

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 subjects withdrew before randomization 12 subjects were excluded due to head circumference >60cm 2 refused randomization 2 subjects were not randomized for an unspecified reason
Period: Overall Study
Arm/Group | 5.5cm Rule Group | F3 Group
Started | 47 | 58
Completed | 41 | 53
Not Completed | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 5.5cm Rule Group | F3 Group | Total
Number analyzed (Participants) | 47 | 58 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (15.8) | 44.7 (15.1) | 43 (15.45)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 30 | 39 | 69
  Male | 16 | 19 | 35
  Female to Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 47 | 57 | 104
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 45 | 56 | 101
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 47 | 58 | 105
Comorbidities [Number; unit: participants]
  Anxiety disorders | 26 | 24 | 50
  OCD | 2 | 4 | 6
  PTSD | 8 | 7 | 15
  ADHD | 3 | 12 | 15
  Borderline Personality Disorder | 7 | 5 | 12
Psychiatric Medications [Count of Participants; unit: Participants] — Number of participants that self-reported medication trials in the reported categories in the current major depressive episode
  Participants
    Antidepressants | 43 | 55 | 98
    Antipsychotics | 18 | 16 | 34
    Benzodiazepines | 17 | 33 | 50
    Stimulants | 9 | 16 | 25
    Mood Stabilizers | 8 | 12 | 20
    Anxiolytics/Hypnotics | 21 | 19 | 40
Number of Medication Trials [Mean (Standard Deviation); unit: medications] — Count of self-reported medication trials that either were not tolerable or did not reduce severity of symptoms in the current major depressive episode
  medications | 10.0 (5.4) | 9.8 (4.9) | 9.9 (5.15)
Patient Health Questionnaire 9-Item Assessment [Mean (Standard Deviation); unit: total score] — This assesses depression severity at baseline. Total scores of 5, 10, 15, and 20 represent markers for mild, moderate, moderately severe, and severe depression, respectively.
  All 9 items are summed to compute a total score, ranging from 0-27. Higher scores indicate more severe self-rated depressive symptoms.
  total score | 18.8 (4.3) | 17.8 (4.9) | 18.3 (4.6)
General Anxiety Disorder 7-Item Assessment [Mean (Standard Deviation); unit: total score] — This assesses anxiety severity as baseline. Scores of 5, 10, and 15 are cut-off points for mild, moderate, and severe anxiety, respectively.
  All 7 items are summed to compute a total score, ranging from 0-21. Higher scores indicate more severe self-rated anxiety symptoms.
  total score | 14.3 (4.7) | 13.5 (5.2) | 13.9 (5.0)
Montgomery-Asberg Depression Rating Scale [Mean (Standard Deviation); unit: total score] — This assesses depression severity at baseline. Scores of 8, 17, and 34 are cut-off points for mild, moderate, severe depression, respectively.
  This 10 item scale is summed to compute a total score, ranging from 0-60. Higher scores indicate more severe clinician-rated depressive symptoms.
  total score | 29.1 (6.9) | 29.8 (5.9) | 29.5 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Patient Health Questionnaire 9-Item Assessment Score
Description: Overall change in total Patient Health Questionnaire 9-Item Assessment score from pre to post-treatment assessment, comparing results of 2 active groups to assess for superiority of one treatment to the other.
  This assessment measures depression severity at baseline. Total scores of 5, 10, 15, and 20 represent markers for mild, moderate, moderately severe, and severe depression, respectively.
  All 9 items are summed to compute a total score, ranging from 0-27. Higher scores indicate more severe self-rated depressive symptoms. Negative change from baseline implies a decrease in depressive symptoms.
Time Frame: Pre-assessment will be obtained within approximately 1 week of starting rTMS. Post-assessment will be obtained immediately following completion of rTMS course, usually 4-6 weeks later.
Measure: Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | 5.5cm Rule Group | F3 Group
Number analyzed (Participants) | 41 | 53
percentage of change from baseline | -38.7 (5.1) | -39.1 (4.7)
Statistical Analysis 1: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures; Test type: Other — comparative effectiveness trial; p = 0.945, t-test, 2 sided

2. Primary Outcome: Percentage Change in Montgomery-Asberg Depression Rating Scale Score
Description: Overall change in total Montgomery-Asberg Depression Rating Scale score from pre to post-treatment assessment, comparing results of 2 active groups to assess for superiority of one treatment to the other.
  This scale assesses depression severity at baseline. Scores of 8, 17, and 34 are cut-off points for mild, moderate, severe depression, respectively.
  This 10 item scale is summed to compute a total score, ranging from 0-60. Higher scores indicate more severe clinician-rated depressive symptoms.
  Negative change from baseline implies a decrease in depressive symptoms.
Time Frame: as for outcome 1
Population: Data reported here includes subjects that had both first and final data point. As such, this group has a smaller sample size.
Measure: Mean (Standard Error); unit: percentage of change from baseline
Arm/Group | 5.5cm Rule Group | F3 Group
Number analyzed (Participants) | 30 | 37
percentage of change from baseline | -39.5 (5.6) | -37.8 (5.6)
Statistical Analysis 1: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures; Test type: Other — comparative effectiveness trial; p = 0.828, t-test, 2 sided

3. Primary Outcome: Percentage Change in General Anxiety Disorder 7-Item Assessment Score
Description: Overall change in total General Anxiety Disorder 7-Item Assessment score from pre to post-treatment assessment, comparing results of 2 active groups to assess for superiority of one treatment to the other.
  This assesses anxiety severity as baseline. Scores of 5, 10, and 15 are cut-off points for mild, moderate, and severe anxiety, respectively.
  All 7 items are summed to compute a total score, ranging from 0-21. Higher scores indicate more severe self-rated anxiety symptoms.
  Negative change from baseline implies a decrease in anxiety symptoms.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Error); unit: percentage change from baseline
Arm/Group | 5.5cm Rule Group | F3 Group
Number analyzed (Participants) | 33 | 43
percentage change from baseline | -33.6 (5.3) | 27.5 (6.9)
Statistical Analysis 1: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures; Test type: Other — comparative effectiveness trial; p = 0.252, t-test, 2 sided

4. Primary Outcome: Response and Remission Rates on Patient Health Questionnaire 9-Item Assessment
Description: Comparison of the response rate (>50% improvement) and remission rate (score <5) for the Patient Health Questionnaire 9-Item Assessment between the 2 groups post-treatment.
Time Frame: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | 5.5cm Rule Group | F3 Group
Number analyzed (Participants) | 41 | 53
percentage of participants
  Responders | 36.6 | 43.4
  Remitters | 22.0 | 20.8
Statistical Analysis 1: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures. A power analysis revealed that a total sample size of 144 would have 80% power when testing for differences between target groups at alpha = 0.05. Accounting for potential attrition, the study conservatively planned to enroll 200 participants, with a planned interim analysis after 100 participants were randomized; Test type: Other; p = 0.505, Chi-squared — p value for response rate
Statistical Analysis 2: Comparison: 5.5cm Rule Group vs F3 Group; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.888, Chi-squared — p value for remission rate

5. Primary Outcome: Response and Remission Rates on Montgomery-Asberg Depression Rating Scale
Description: Comparison of the response rate (>50% improvement) and remission rate (score <10) for the MADRS between the 2 groups post-treatment.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | 5.5cm Rule Group | F3 Group
Number analyzed (Participants) | 30 | 37
percentage of participants
  Responders | 43.3 | 43.2
  Remitters | 20.0 | 18.9
Statistical Analysis 1: Comparison: 5.5cm Rule Group vs F3 Group; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.994, Chi-squared; p value for response rates
Statistical Analysis 2: Comparison: 5.5cm Rule Group vs F3 Group; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.911, Chi-squared; p value for remission rates

6. Primary Outcome: Response Rates on General Anxiety Disorder 7-Item Assessment
Description: Comparison of the response rate (>50% improvement) for the General Anxiety Disorder 7-Item Assessment between the 2 groups post-treatment.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | 5.5cm Rule Group | F3 Group
Number analyzed (Participants) | 33 | 43
percentage of participants | 27.3 | 30.2
Statistical Analysis 1: Comparison: 5.5cm Rule Group vs F3 Group; [analysis description as in outcome 4, analysis 1]; Test type: Other; p = 0.778, t-test, 2 sided

7. Secondary Outcome: Montreal Cognitive Assessment Score Changes
Description: Change in Montreal Cognitive Assessment scores from baseline to final timepoint. Reported here as the mean difference in total Montreal Cognitive Assessment score from baseline to endpoint.
  Montreal Cognitive Assessment is used a screen for cognitive impairment, calculated by adding the points from each task, which range from 0-30.
  Higher scores indicate little to no cognitive impairment 26 or above: Normal cognition 18-25: Mild cognitive impairment 10-17: Moderate cognitive impairment Fewer than 10: Severe cognitive impairment
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 5.5cm Rule Group | F3 Group
Number analyzed (Participants) | 29 | 36
score on a scale | .59 (2.3) | .56 (1.8)
Statistical Analysis 1: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures; Test type: Other — comparative effectiveness trial; p = .951, t-test, 2 sided

8. Secondary Outcome: Emotion Measures
Description: T Score Changes in National Institutes of Health Toolbox Emotional Battery A T score of 50 corresponds to the population mean. Scores may range from 20-80 with a standard deviation of 10. Higher T scores indicate a higher endorsement of each domain. Here, we present changes in mean score from pre-treatment to post-treatment. In that way, a positive value represents a decrease in average T score, and vice versa.
Time Frame: as for outcome 1
Population: Only a subset of participants completed this task, so total sample size is much smaller.
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | 5.5cm Rule Group | F3 Group
Number analyzed (Participants) | 17 | 23
T Score
  Positive Affect | -7.2 (9.4) | -10.4 (8.9)
  General Life Satisfaction | -2.7 (7.1) | -9.2 (9.6)
  Meaning & Purpose | -4.5 (8.0) | -6.7 (9.5)
  Emotional Support | -0.2 (8.7) | -6.9 (9.0)
  Instrumental Support | 3.9 (9.4) | -5 (10.1)
  Friendship | 0.1 (5.3) | -5.4 (7.5)
  Loneliness | 3.2 (11.1) | 5.8 (8.5)
  Perceived Rejection | -1.3 (10.5) | 4.7 (9.3)
  Perceived Hostility | 1.8 (8.1) | 4.3 (9.1)
  Self-Efficacy | -1.6 (6.3) | -3.2 (7.6)
  Perceived Stress | 4.6 (12.0) | 7.6 (8.8)
  Fear-Affect | 4.9 (6.7) | 6.9 (8.6)
  Fear-Somatic Arousal | -1.1 (10.9) | 4.4 (9.4)
  Sadness | 7.0 (14.5) | 13.2 (10.9)
  Anger-Affect | 6.5 (11.1) | 6.3 (11.6)
  Anger-Hostility | 2.1 (12.2) | 2.7 (8.8)
  Anger-Physical Aggression | 3.4 (9.2) | -0.6 (4.9)
  Negative Affect | 6.1 (11.7) | 8.7 (7.8)
  Social Satisfaction | 0.2 (8.5) | -7.2 (9.4)
  Psychological Well Being | -5.6 (8.2) | -10.2 (9.1)
Statistical Analysis 1: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures. Results below are for the subscale, Positive Affect; Test type: Other — comparative effectiveness trial; p = .278, t-test, 2 sided
Statistical Analysis 2: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures. Results below are for the subscale, General Life Satisfaction; Test type: Other — comparative effectiveness trial; p = .024, t-test, 2 sided
Statistical Analysis 3: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures. Results below are for the subscale, Meaning & Purpose; Test type: Other — comparative effectiveness trial; p = .439, t-test, 2 sided
Statistical Analysis 4: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures. Results below are for the subscale, Emotional Support; Test type: Other — comparative effectiveness trial; p = .025, t-test, 2 sided
Statistical Analysis 5: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures. Results below are for the subscale, Instrumental Support; Test type: Other — comparative effectiveness trial; p = .007, t-test, 2 sided
Statistical Analysis 6: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures. Results below are for the subscale, Friendship; Test type: Other — comparative effectiveness trial; p = .014, t-test, 2 sided
Statistical Analysis 7: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures. Results below are for the subscale, Loneliness; Test type: Other — comparative effectiveness trial; p = .398, t-test, 2 sided
Statistical Analysis 8: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures. Results below are for the subscale, Perceived Rejection; Test type: Other — comparative effectiveness trial; p = .064, t-test, 2 sided
Statistical Analysis 9: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures. Results below are for the subscale, Perceived Hostility; Test type: Other — comparative effectiveness trial; p = .368, t-test, 2 sided
Statistical Analysis 10: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures. Results below are for the subscale, Self-Efficacy; Test type: Other — comparative effectiveness trial; p = .504, t-test, 2 sided
Statistical Analysis 11: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures. Results below are for the subscale, Perceived Stress; Test type: Other — comparative effectiveness trial; p = .371, t-test, 2 sided
Statistical Analysis 12: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures. Results below are for the subscale, Fear-Affect; Test type: Other — comparative effectiveness trial; p = .438, t-test, 2 sided
Statistical Analysis 13: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures. Results below are for the subscale, Fear-Somatic Arousal; Test type: Other — comparative effectiveness trial; p = .096, t-test, 2 sided
Statistical Analysis 14: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures. Results below are for the subscale, Sadness; Test type: Other — comparative effectiveness trial; p = .132, t-test, 2 sided
Statistical Analysis 15: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures. Results below are for the subscale, Anger-Affect; Test type: Other — comparative effectiveness trial; p = .951, t-test, 2 sided
Statistical Analysis 16: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures. Results below are for the subscale, Anger-Hostility; Test type: Other — comparative effectiveness trial; p = .852, t-test, 2 sided
Statistical Analysis 17: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures. Results below are for the subscale, Anger-Physical Aggression; Test type: Other — comparative effectiveness trial; p = .083, t-test, 2 sided
Statistical Analysis 18: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures. Results below are for the subscale, Negative Affect; Test type: Other — comparative effectiveness trial; p = .391, t-test, 2 sided
Statistical Analysis 19: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures. Results below are for the subscale, Social Satisfaction; Test type: Other — comparative effectiveness trial; p = .014, t-test, 2 sided
Statistical Analysis 20: Comparison: 5.5cm Rule Group vs F3 Group; The null hypothesis of this study was that there would be no differences between targets across all measures. Results below are for the subscale, Psychological Well Being; Test type: Other — comparative effectiveness trial; p = .109, t-test, 2 sided

9. Post Hoc Outcome: Patient Health Questionnaire 9-Item Assessment Linear Mixed Effects Model
Description: An exploratory analysis to investigate between-group differences in trajectory of improvement as measured by group by time interactions.
  This assessment measures depression severity at baseline. Total scores of 5, 10, 15, and 20 represent markers for mild, moderate, moderately severe, and severe depression, respectively.
  All 9 items are summed to compute a total score, ranging from 0-27. Higher scores indicate more severe self-rated depressive symptoms. Negative change from baseline implies a decrease in depressive symptoms.
Time Frame: Baseline to Weeks 1 through 6, assessed weekly
Population: All randomized participants were included in this analysis. Weekly timepoints have different ns due to dropouts and/or missing data.
Measure: Mean (Standard Deviation); unit: mean PHQ-9 total score
Arm/Group | 5.5cm Rule Group | F3 Group
Number analyzed (Participants) | 46 | 58
mean PHQ-9 total score
  First Visit | 18.8 (4.3) | 17.8 (4.9)
  Week 1: number analyzed (Participants) | 44 | 57
  Week 1 | 15.7 (6.2) | 16.2 (5.9)
  Week 2: number analyzed (Participants) | 44 | 55
  Week 2 | 14.6 (6.3) | 14.4 (6.3)
  Week 3: number analyzed (Participants) | 43 | 54
  Week 3 | 14.2 (6.7) | 12.6 (6.4)
  Week 4: number analyzed (Participants) | 41 | 53
  Week 4 | 13.2 (6.3) | 13.0 (6.5)
  Week 5: number analyzed (Participants) | 42 | 51
  Week 5 | 12.5 (6.3) | 11.8 (7.1)
  Week 6: number analyzed (Participants) | 37 | 51
  Week 6 | 10.7 (6.7) | 11.2 (7.5)
Statistical Analysis 1: Comparison: 5.5cm Rule Group vs F3 Group; Test type: Superiority; p = 0.231, Mixed Models Analysis — Week 6 timepoint p-value listed above; Other timepoint p-values below: First Visit p = 0.875 Week 1 p = 0.084 Week 2 p = 0.277 Week 3 p = 0.686 Week 4 p = 0.369 Week 5 p = 0.806

10. Post Hoc Outcome: Montgomery-Asberg Depression Rating Scale Linear Mixed Effects Model
Description: An exploratory analysis to investigate between-group differences in trajectory of improvement as measured by group by time interactions.
  This scale assesses depression severity at baseline. Scores of 8, 17, and 34 are cut-off points for mild, moderate, severe depression, respectively.
  This 10 item scale is summed to compute a total score, ranging from 0-60. Higher scores indicate more severe clinician-rated depressive symptoms.
  Negative change from baseline implies a decrease in depressive symptoms.
Time Frame: Baseline to biweekly timepoints
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mean MADRS total score
Arm/Group | 5.5cm Rule Group | F3 Group
Number analyzed (Participants) | 42 | 57
mean MADRS total score
  Evaluation | 29.1 (6.9) | 29.8 (5.9)
  Week 2-3 Follow-up: number analyzed (Participants) | 40 | 45
  Week 2-3 Follow-up | 24.2 (8.1) | 22.0 (7.2)
  Week 4-5 Follow-up: number analyzed (Participants) | 37 | 42
  Week 4-5 Follow-up | 18.4 (9.3) | 19.6 (8.7)
  Week 6-7 Follow-up: number analyzed (Participants) | 35 | 46
  Week 6-7 Follow-up | 15.3 (8.8) | 16.4 (9.7)
Statistical Analysis 1: Comparison: 5.5cm Rule Group vs F3 Group; Test type: Superiority; p = 0.963, Mixed Models Analysis — Week 6-7 Follow-up p-value listed above; Other timepoint p-values below: Evaluation p = 0.570 Week 2-3 Follow-up p = 0.063 Week 4-5 Follow-up p = 0.792

11. Post Hoc Outcome: General Anxiety Disorder 7-Item Assessment Linear Mixed Effects Model
Description: An exploratory analysis to investigate between-group differences in trajectory of improvement as measured by group by time interactions.
  This assesses anxiety severity as baseline. Scores of 5, 10, and 15 are cut-off points for mild, moderate, and severe anxiety, respectively.
  All 7 items are summed to compute a total score, ranging from 0-21. Higher scores indicate more severe self-rated anxiety symptoms.
  Negative change from baseline implies a decrease in anxiety symptoms.
Time Frame: Baseline to weekly timepoints
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: mean GAD-7 total score
Arm/Group | 5.5cm Rule Group | F3 Group
Number analyzed (Participants) | 37 | 48
mean GAD-7 total score
  First Visit | 14.3 (4.7) | 13.5 (5.2)
  Week 1: number analyzed (Participants) | 36 | 46
  Week 1 | 12.3 (5.1) | 12.6 (5.2)
  Week 2: number analyzed (Participants) | 36 | 44
  Week 2 | 10.9 (5.4) | 11.3 (5.7)
  Week 3: number analyzed (Participants) | 34 | 44
  Week 3 | 10.7 (5.7) | 10.8 (5.6)
  Week 4: number analyzed (Participants) | 33 | 43
  Week 4 | 9.7 (4.9) | 10.6 (6.4)
  Week 5: number analyzed (Participants) | 33 | 42
  Week 5 | 9.6 (5.5) | 10.0 (6.5)
  Week 6: number analyzed (Participants) | 30 | 42
  Week 6 | 9.0 (5.6) | 10.0 (6.6)
Statistical Analysis 1: Comparison: 5.5cm Rule Group vs F3 Group; Test type: Superiority; p = 0.051, Mixed Models Analysis — Week 6 timepoint p-value listed above; Other timepoint p-values below: First Visit p = 0.772 Week 1 p = 0.194 Week 2 p = 0.127 Week 3 p = 0.196 Week 4 p = 0.079 Week 5 p = 0.187

ADVERSE EVENTS:
Time Frame: During the course of TMS treatment (approx. 4-6 weeks)
Arm/Group | 5.5cm Rule Group | F3 Group
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/58
Other Adverse Events (participants affected / at risk) | 0/47 | 0/58

LIMITATIONS AND CAVEATS:
* The study study sample included many people with significant psychiatric comorbidities, was predominately white and non-Hispanic, and did not standardize or control medication changes.
* Subjects were not randomized into iTBS or 10 Hz.
* There was lack of assessment of blinding.
* This study excluded participants with a head circumference >60 cm.
* Due to the naturalistic sample, a cut-off of having received at least 20 treatments was used for inclusion in the primary analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/70/NCT03378570/Prot_002.pdf
  • Statistical Analysis Plan (2019-08-22): https://cdn.clinicaltrials.gov/large-docs/70/NCT03378570/SAP_003.pdf